CLINICAL TRIAL: NCT05254977
Title: Data Collection for Post Vaccination Adverse Events in Covid-19 Vaccine Recipients in District Bahawalpur A Multi-center Observational Study
Brief Title: Post Vaccination Adverse Events in Covid-19 Vaccine Recipients
Status: Completed | Type: Observational
Sponsor: Islamia University of Bahawalpur (Other)
Collaborators: District Health Authority (DHA) Bahawalpur District Bahawalpur, Government of Punjab. (Unknown)
Responsible Party: Principal Investigator, Hafiz Abdul Sattar Hashmi, Lecturer, Islamia University of Bahawalpur
Other Study IDs: UCCM/2022/Covid-19/01
Record Dates: First submitted 2022-02-19; First posted 2022-02-24 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Vaccination; Vaccine Adverse Reaction
Keywords: Covid-19 Vaccination, Inactivated Vaccine, RNA vaccine
MeSH Terms: interventions — Reference Standards

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (28):
- B.V. HOSPITAL: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- Baldia Hall Yazman: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- CIVIL HOSPITAL Bahahwalpur: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- DDHO KPT: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- Govt Girls Elementry School: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- Govt Higher Secondary School: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- Govt Sadiq Higher Secondary School: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- Govt TibIA College Bahawalpur: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- CEO Office DHA BWP: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- Papulation Welfare office APE: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Ballah Jhulan: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Channi Goth: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Choona wala: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Dera Bakha: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Headrajkan: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Khanqah sharif: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Khutri Banglow: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Kud Wala: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Lal Sohanra: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Mubarkpur: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Qaimpur: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- RHC Uch Sharif: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- Special Education Degree Colage: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- THQ HOSPITAL, AHMADPUR: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- THQ HOSPITAL, HASILPUR.: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- THQ KHAIR PUR TAMEWALI: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- THQ YAZMAN: Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation
- TMA Office Hasilpur (NEW): Local population in surrounding premises of site
  Interventions: Drug: Standard Preparation

INTERVENTIONS:
Drug: Standard Preparation — Any kind of intervention received to reduce adverse effects

SUMMARY:
Covid-19 pandemic is caused by Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-Cov-2) since its outbreak 2019. Protection against Covid-19 can be achieved through global immunization. Various vaccines for SARS-Cov-2 has been registered and approved for administration in humans. It is important to understand the safety and efficacy of vaccines during robust research to develop global immunity against SARS-Cov-2. This study aimed to collect data on post vaccination adverse events in regional population of District Bahawalpur.

DETAILED DESCRIPTION:
Bahawalpur District of Punjab province has population of 3.998 million and among these 2.6 million above 12 years of age are eligible for vaccination against SARS-Cov-2. 28 centers were established for vaccination within the districts at designated sites for Covid-19 vaccination. 87% targeted population has been vaccinated till 15th February 2022. Investigators designed this study to collect and evaluate data on adverse effects after vaccination of Covid-19. Investigators aimed to collect information through interviewing participants in general places of designated sites of vaccination centers established in District Bahawalpur. History will be recorded from participants and in case of adverse events detailed available history will be recorded including following adverse effects from available records on following.

* Cardiovascular adverse effects
* Cerebrospinal adverse events
* Respiratory disturbances
* Hepatobiliary disorders
* Urogenital adverse effects
* Musculoskeletal adverse effect
* Psychological diseases
* Blood biomarkers changes
* Autoimmune adverse events
* Allergic reactions and hypersensitivity Collected data will be summarized to get percentage of adverse effects in general population. Recorded adverse events will be assessed for their frequency in participants and association with vaccination will be assessed through employing statistical methods. Subsequent information on handling of adverse events will be recorded including
* Nature of adverse event
* Hospitalization and severity of adverse events
* Mortality / morbidity caused by vaccination
* Days of hospitalization
* Changes in Blood biomarkers
* Interventions adopted for adverse events
* Diseased period
* Covid-19 infection positivity through RT-PCR / imaging for round glass opacities / Covid-19 changes Overall efficacy and safety of vaccination will be assessed through collected data.

ELIGIBILITY:
Inclusion Criteria:

Age >12 year Vaccinated (Single Dose, Double Dose, Booster Dose) Clinical diagnosis of Allergic reactions and hypersentivity, Cardiovascular diseases Musculoskeletal diseases Respiratory disease Immunological disease Kidney diseases

Exclusion Criteria:

Age <12 years of age Not vaccinated History of disease before vaccination

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population above age of 12 years will be eligible to collection information on adverse effects of SARS-Cov-2 vaccination
Sampling Method: Probability Sample
Enrollment: 3515 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Allergic reactions and hypersensitivity | 1st January 2021 to 31st December 2021
  Questionnaire for Allergic reaction at injection site or generalized allergic responses excluding previously known disease
Cardiovascular Diseases | 1st January 2021 to 31st December 2021
  Questionnaire for Post Vaccination adverse development of Hypertension, heart diseases, vascular diseases excluding previously known disease
Respiratory disorders and Respiratory hypersensitivity | 1st January 2021 to 31st December 2021
  Questionnaire for Cough, dyspnea, Tachypnea, Asthma, Rhinitis, excluding previously known disease
Urologic Diseases | 1st January 2021 to 31st December 2021
  Questionnaire for Kidney diseases, Urinary tract infection, Urolithiasis excluding previously known disease
Immune system disorders | 1st January 2021 to 31st December 2021
  Questionnaire for Autoimmune diseases, Erythroblastosis, Glomerulonephritis, thrombocytopenia, Autoimmune Lymphoproliferative Syndrome excluding previously known disease
Musculoskeletal diseases | 1st January 2021 to 31st December 2021
  Questionnaire for fatigue syndrome, muscle weakness, muscle spasticity, muscle rigidity, Musculoskeletal pain, myalgia, osteoarthritis, Myositis excluding previously known disease

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Abdul Sattar, M.Phil, Principal Investigator — Lecturer
Locations (1):
- University College of Conventional Medicine, Bahawalpur, Punajb, Pakistan

IPD SHARING:
Plan to Share IPD: No